CLINICAL TRIAL: NCT05240261
Title: Effects of Sleep Disorders and Sedative-hypnotic Medications on Health-related Quality of Life in Chronic Kidney Disease Patients
Brief Title: Sleep Disorders in Chronic Kidney Disease Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mona Abd Ellatif Aly Ismael, specialist of nephrology., Assiut University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Chronic kidney disease (CKD)
Record Dates: First submitted 2022-01-02; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESRAD on regular haemodialysis (Other): 30 ESRD Patients with sleep < 6 hours on regular haemodialysis . Before and after taking medications for 3 month.
  Interventions: Drug: Quetiapine
- CKD patients (predialydsis) (Other): 30 CKD Patients (predialysis) with sleep < 6 hours . Before and after taking medications for 3 month.
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — Quetiapine 25 mg / day

SUMMARY:
1. Asses sleep disorders in CKD patients and those on haemodialysis and related complications ( uncontrolled blood pressure,glomerular filtration rate (GFR) ,proteinuria and psychological disturbance)
2. Asses effect of hypnotics or sedations for 3 month in improvement those complications after taking treatment .

DETAILED DESCRIPTION:
Sleep disorders are prevalent in patients with chronic kidney disease (CKD) in particular those with end stage renal disease (ESRD). It has been reported that 80% of ESRD patients receiving dialysis report sleep complaints, with daytime sleepiness to be the most common reported symptom. The reason for increased rates of sleep related issues and disorders in this population is likely multifactorial.

Although it is commonly accepted that patients with CKD experience poor sleep quality, not much is known about the physiological mechanisms underlying this phenomenon. Patients with CKD often exhibit sympatho-vagal imbalance due to baroreceptor reflex function impairment in which there is hyperactivity of the sympathetic nervous system and decreased vagal tone. In healthy individuals, sleep is accompanied by a decrease in sympathetic activity and an increase in vagal tone that leads to a nocturnal dipping of blood pressure. However, patients who have sleep disorders resulting in hypoxemia and sleep fragmentation have been shown to have increased sympathetic nervous system stimulation and decreased parasympathetic activity, which results in a reduced fall in nocturnal blood pressure.

In patients with ESRD, the identification, diagnosis and treatment of sleep disorders is complicated by the overlapping presentation with CKD and other commonly comorbid conditions. One approach to conceptualizing this relationship is to consider sleep disorders as secondary or end product of multiple concurrent and interactive processes. Such processes include psychological disorders (depression, anxiety), lifestyle factors (coffee/nicotine use, sleep hygiene), treatment-related factors (timing of dialysis, daytime napping, production of cytokines, thermoregulatory changes, dialysis disequilibrium syndrome, disruptions in circadian rhythm, medication side effects) as well as intrinsic, ESRD-specific factors (anemia/obstructive sleep apnea (OSA) and other comorbidities, uremia, overall all health and quality of life, alterations in neurotransmitter production).

A poor sleep profile is associated with increased risk of CKD development. Therefore, sleep duration and quality should be considered when developing strategies to improve sleep and thus prevent CKD.

Poor sleep quality, which is commonly found in pre-dialysis CKD patients, is an independent factor associated with cardiovascular damage in CKD patients.

Both short and long sleep durations are significantly associated with CKD and proteinuria. Some findings suggest curvilinear dose-response associations of sleep duration with CKD and proteinuria.

Optimizing sleep quality and duration to >6 h/night improved BP control and was associated with a significant delta change in systolic blood pressure (SBP) within 3 months of follow-up. Physicians should obtain a sleep history in patients with CKD who present with resistant hypertension.

Poor sleep quality is prevalent in patients on maintenance haemodialysis, and is associated with increased daytime sleepiness. Depression further compounds this relationship, and is significantly associated with increased daytime sleepiness and restless leg syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 1.patients are between ages 18 and 60 with chronic kidney disease (CKD)( stage III-V) and ESRD Patients on regular haemodialysis > 6 months.and time of start session of dialysis at 5 pm , thrice weekly .

  2. Random urine albumin/creatinine ratio of 30 mcg/day or greater (protein in the urine) 3. Patients have ability to complete a sleep survey and must be able to swallow tablets.

  4. Patients with compensated heart and liver disease. 5. Not on antipsychotic drugs.

Exclusion Criteria:

1. Patients with history of psychosis.
2. Patients with decompensated heart or liver disease.
3. Patients with diabetes , autoimmune ,thyroid or neurological disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
1- change in Blood pressure measurement . | 3 months
  follow up blood pressure ( millimeters of mercury (mm/hg)
The Quality of Life Scale (QOLS) | 3 months
  Scores can range from 16 to 112. higher scores indicate better life quality.
Pittsburgh Sleep Quality Index score (PSQI S). | 3 months
  Scale 0-21, higher scores indicate worse sleep quality.

SECONDARY OUTCOMES:
change in Estimated Glomerular filteration rate. | 3 month
proteinuria | 3 months

REFERENCES:
- [Background] Zhang J, Wang C, Gong W, Peng H, Tang Y, Li CC, Zhao W, Ye Z, Lou T. Association between sleep quality and cardiovascular damage in pre-dialysis patients with chronic kidney disease. BMC Nephrol. 2014 Aug 12;15:131. doi: 10.1186/1471-2369-15-131. PMID 25117823
- [Background] Pengo MF, Ioratti D, Bisogni V, Ravarotto V, Rossi B, Bonfante L, Simioni F, Nalesso F, Maiolino G, Calo LA. In Patients with Chronic Kidney Disease Short Term Blood Pressure Variability is Associated with the Presence and Severity of Sleep Disorders. Kidney Blood Press Res. 2017;42(5):804-815. doi: 10.1159/000484357. Epub 2017 Nov 28. PMID 29212081
- [Background] Parvan K, Lakdizaji S, Roshangar F, Mostofi M. Quality of sleep and its relationship to quality of life in hemodialysis patients. J Caring Sci. 2013 Nov 30;2(4):295-304. doi: 10.5681/jcs.2013.035. eCollection 2013 Dec. PMID 25276738
- [Background] Hao Q, Xie M, Zhu L, Dou Y, Dai M, Wu Y, Tang X, Wang Q. Association of sleep duration with chronic kidney disease and proteinuria in adults: a systematic review and dose-response meta-analysis. Int Urol Nephrol. 2020 Jul;52(7):1305-1320. doi: 10.1007/s11255-020-02488-w. Epub 2020 May 16. PMID 32418007